CLINICAL TRIAL: NCT00488267
Title: A Randomized, Double-Blind, 12-Week Study to Evaluate the Efficacy of ThermoProfen™ in the Treatment of Patients With Mild to Moderate Pain Associated With Osteoarthritis of the Knee (ZMK-301)
Brief Title: Efficacy of ThermoProfen in Patients With Mild to Moderate Pain Associated With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZMK-301
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Thermoprofen (Experimental): ThermoProfen™ (ketoprofen matrix/Controlled Heat Assisted Drug Delivery [CHADD™] patch)
  Interventions: Drug: ThermoProfen™ (Matrix Transdermal Ketoprofen/CHADD™ System)
- Placebo Matrix (Placebo Comparator): Placebo matrix with CHADD patch.
  Interventions: Drug: Placebo Matrix/CHADD Patch
- Ketoprofen matrix/placebo CHADD (Placebo Comparator): Ketoprofen matrix with placebo CHADD patch (no heat)
  Interventions: Drug: Ketoprofen matrix/placebo CHADD Patch

INTERVENTIONS:
Drug: ThermoProfen™ (Matrix Transdermal Ketoprofen/CHADD™ System) — Transdermal patch applied to the knee for 12 hours daily.
  Other Names: Matrix Transdermal Ketoprofen CHADD System
  Arms: Thermoprofen
Drug: Placebo Matrix/CHADD Patch — Transdermal patch applied to the knee for 12 hours daily.
  Other Names: Placebo patch with heating system
  Arms: Placebo Matrix
Drug: Ketoprofen matrix/placebo CHADD Patch — Transdermal knee applied to the knee for 12 hours daily.
  Other Names: ketoprofen matrix with no heat
  Arms: Ketoprofen matrix/placebo CHADD

SUMMARY:
ThermoProfen is a transdermal ketoprofen patch that is integrated with a long-lasting CHADD (Controlled Heat-Assisted Drug Delivery) unit for the treatment of chronic pain associated with osteoarthritis. This study will evaluate ThermoProfen for the treatment of mild to moderate pain associated with osteoarthritis of the knee in adults.

DETAILED DESCRIPTION:
The primary objective of the study is to compare the efficacy of ThermoProfen™ against two other experimental treatments.

The treatment may be ThermoProfen (Matrix Transdermal Ketoprofen Patch) or a patch that may or may not include ketoprofen and that may or may not provide heat.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 through 75 years of age
* Patient has radiographic evidence of osteoarthritis of the target knee obtained within the past year.

Exclusion Criteria:

* Patient has a known allergy to nonsteroidal anti-inflammatory drugs (NSAIDs, including aspirin).
* Patient has asthma that has been induced or made worse by the use of aspirin or NSAIDs.
* Patient has a relevant history of serious gastrointestinal disease.
* Patient, if female, is pregnant or breastfeeding or is of childbearing potential and not practicing adequate birth control.
* Patient is taking warfarin, heparin, or low molecular weight heparin.
* Patient has received oral, intramuscular, intravenous, intra-articular, or soft-tissue administration of steroids within 1 month of study enrollment (or within 2 months, if in the target joint).
* Patient has received intra-articular visco-supplementation (in target joint) within 6 months of study enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the change from baseline in the Visual Analog Scale score for the average pain during the previous 24 hours. | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in Visual Analog Scale score for worst pain during the previous 24 hours, amount of rescue medication used to treat the target joint per day, and the patient global impression of change in the Likert Scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — ZARS Pharma
Locations (36):
- United States (36):
  - Peoria, Arizona
  - Anaheim, California
  - Buena Park, California
  - San Diego, California
  - Westlake Village, California
  - Hamden, Connecticut
  - Milford, Connecticut
  - Clearwater, Florida
  - Jupiter, Florida
  - Pembroke Pines, Florida
  - South Miami, Florida
  - Tampa, Florida
  - Boise, Idaho
  - Springfield, Illinois
  - Evansville, Indiana
  - Overland Park, Kansas
  - Baltimore, Maryland
  - Wheaton, Maryland
  - Lansing, Michigan
  - Kansas City, Missouri
  - Mercerville, New Jersey
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Duncansville, Pennsylvania
  - Erie, Pennsylvania
  - Mechanicsburg, Pennsylvania
  - Anderson, South Carolina
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Spokane, Washington
  - Tacoma, Washington